CLINICAL TRIAL: NCT06584799
Title: Comparative Assessment of the Efficacy and Safety of Venoactive Drug Treatment of Pelvic Venous Disorders
Brief Title: Venoactive Drug Treatment of Pelvic Venous Disorders
Acronym: VENOTREAT
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Pirogov Russian National Research Medical University (Other)
Responsible Party: Principal Investigator, Sergey Gavrilov, MD, PhD, Professor, Pirogov Russian National Research Medical University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 20452024
Record Dates: First submitted 2024-08-29; First posted 2024-09-05 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Pelvic Venous Disorders
Keywords: pelvic venous disorders; chronic pelvic pain; venoactive drug therapy; pelvic pain
MeSH Terms: conditions — Pelvic Pain

STUDY DESIGN:
Intervention Model Description: Clinical trials with a single arm. The study will include 150 consecutive female patients with symptomatic PeVD. All patients will undergo a clinical examination, transabdominal and transvaginal DUS of the pelvic veins to verify the diagnosis and to determine the diameters of the pelvic veins and the duration of reflux in them. The CPP intensity will be assessed using a visual analogue scale (VAS). For randomization procedure, the sealed envelope principle will be used. Three groups of 50 patients each will be formed depending on the recommended VAD usage: group 1 (n=50) with MPFF1000; group 2 (n=50) with Diosmin 600; and group 3 (n=50) with Hesperidin + Diosmin 1000. After the start of VAD intake, the patients will be self-rating the pain intensity on VAS on the weekly basis. Based on the repeated examination data and the VAS results, a comparative analysis of the clinical efficacy of VADs will be carried out.
Masking Description: Sealed envelope principle
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Active Comparator): Group will include 50 patients, which will be treated by MPFF 1000 mg once daily for 2 months
  Interventions: Drug: Micronized purified flavonoid fraction
- Group 2 (Active Comparator): Group will include 50 patients which will be treated by Diosmin 600 mg once daily for 2 months
  Interventions: Drug: Diosmin 600
- Group 3 (Active Comparator): Group will include 50 patients which will be treated by combination Hespiridin+Diosmin 1000 mg once daily for 2 months
  Interventions: Drug: Hesperidin+Diosmin combination 1000

INTERVENTIONS:
Drug: Micronized purified flavonoid fraction — Micronized purified flavonoid fraction (MPFF) 1000. Active substance: micronized purified flavonoid fraction (diosmin+flavonoids expressed as hesperidin). MPFF is a venotonic agent that also has angioprotective properties. It reduces venous distensibility and blood stasis, capillary permeability, and increases capillary resistance.
  MOFF 1000 dosing regimen is 1000 mg once daily for 2 months.
  Arms: Group 1
Drug: Diosmin 600 — Venotonic action: the drug reduces venous distensibility, increases venous tone, reduces blood stasis, and enhances the vasoconstrictor effect of epinephrine and norepinephrine. The optimal daily dose of diosmin 600 for obtaining venotonic effect is 600 mg.
  Arms: Group 2
Drug: Hesperidin+Diosmin combination 1000 — A venotonic agent that also has angioprotective properties. It reduces venous distensibility and blood stasis, reduces capillary permeability and increases their resistance.
  Hesperidin+Diosmin combination 1000 dosing regimen is 1000 mg once daily for 2 months
  Arms: Group 3

SUMMARY:
Venoactive drug (VAD) therapy is one of the most effective methods of treating chronic venous diseases (CVD). Numerous studies have proven its high efficacy in relieving symptoms of CVD, such as leg pain and swelling, leg heaviness and fatigue. Pelvic venous disorders (PeVDs) represent a group of pathological conditions including varicose veins of the pelvis and vulva, and compression stenoses of the left renal and common iliac veins. Although PeVDs are associated with venous lesions of the pelvis and retroperitoneum and have specific clinical manifestations, they are one of the forms of CVD and constitute a separate cohort. A number of studies on the VAD usage in PeVD indicate the wide possibilities of this type of treatment in eliminating chronic pelvic pain (CPP), the most dramatic symptom of PeVD, which is the main cause of disability and decreased quality of life, social and daily activity in women with PeVD. Currently, a variety of VADs are presented on the pharmaceutical market, which, according to the product labels, provide effects not only on the venous outflow from the lower extremities, but also on venous hemodynamics in the pelvis. At the same time, a literature analysis shows that micronized purified flavonoid fraction (MPFF) has the greatest evidence base obtained in the efficacy and safety studies of VADs in PeVD. Nevertheless, patients are rarely interested in the scientific dossier of drugs, and in the real practice the patients with PeVD and CPP most often ask: "What is the best drug to use for the CPP relief?" This is quite understandable, as it is CPP in PeVD that results not only in disability, but also in family conflicts, psycho-emotional stress and depressive states. In this regard, patients seek to get rid of pain as soon as possible and strive to use the most effective drug. An extensive scientific base of comparative studies on the use of various VADs in patients with CVD and PeVD has been accumulated to date. However, the literature is lack of any data on the comparative efficacy and safety of VADs in the treatment of patients with PeVD. This, in turn, makes not possible for doctors and patients to choose the optimal and most effective drug based on the objective research data. All the above has predetermined the purpose of the planned study as evaluating the efficacy and safety of different VADs in the treatment of female patients with PeVD.

DETAILED DESCRIPTION:
Study objectives:

* To evaluate the efficacy of diosmin-containing VADs in the CPP relief in female patients with PeVD;
* To evaluate the safety (by the number of side effects and adverse events) of diosmin-containing VADs in female patients with PeVD;
* To compare the efficacy and safety of treatment with different diosmin-containing VADs;
* To evaluate the patients' adherence to the different recommended diosmin-containing VADs in female patients with PeVD.

Patients and methods: A total of 150 female patients of reproductive age with symptomatic PeVD and without any other diseases accompanied by CPP are planned for the inclusion in the study.

Clinical study: All patients will be examined by an investigating physician. Complaints, medical history, and physical examination results will be recorded in the individual patient's case report form (CRF). The severity of CPP will be assessed using a 10-score visual analogue scale (VAS) before treatment and then weekly for 2 months of treatment with VAD.

Diagnostic methods:

All patients will undergo transabdominal and transvaginal duplex ultrasound study (DUS) of the pelvic veins.

Treatment methods: the following VADs will be used as the study drugs.

1. Micronized purified flavonoid fraction 1000. Manufacturer: SERVIER RUS, LLC (Russia). Active substance: micronized purified flavonoid fraction (diosmin+flavonoids expressed as hesperidin).

   Micronized purified flavonoid fraction (MPFF) is a venotonic agent that also has angioprotective properties. It reduces venous distensibility and blood stasis, capillary permeability, and increases capillary resistance. The results of clinical studies confirm the pharmacological activity of drugs containing this active substance in relation to the parameters of venous hemodynamics. MPFF improves venous tone: a reduction in venous emptying time has been shown by venous occlusion plethysmography. In patients with signs of severe microcirculatory disorders the treatment with drugs containing this active substance is associated with a statistically significant (as compared to placebo) improvement in the capillary resistance, as has been shown by angiostereometry. The drug also has a proven efficacy in the treatment of CVD of the lower extremities (Source: https://www.vidal.ru/drugs/detralex__38634; accessed: September 4, 2023).

   MPFF 1000 dosing regimen is 1000 mg once daily for 2 months.
2. Diosmin 600. Manufacturer: INNOTHERA CHOUZY (France). Active substance: diosmin.

   Venotonic action: the drug reduces venous distensibility, increases venous tone, reduces blood stasis, and enhances the vasoconstrictor effect of epinephrine and norepinephrine. The optimal daily dose of diosmin for obtaining venotonic effect is 600 mg.

   Angioprotective action: the drug improves microcirculation, increases capillary resistance, and reduces capillary permeability. Effect on the lymphatic system: the drug improves lymphatic drainage, increases the tone and frequency of contraction of lymphatic capillaries, increases their functional density, and reduces lymphatic pressure. It has an anti-edematous effect, reduces symptoms of inflammation (dose-dependent effect), reduces adhesion of leukocytes to the venous wall and their migration into paravasal tissues, and improves oxygen diffusion and perfusion in tissues. The drug hinders the production of free radicals and synthesis of prostaglandins and thromboxane. A double-blind, placebo-controlled study using Duplex ultrasound has confirmed that the drug reduces the mean venous pressure in the system of superficial and deep veins of the lower extremities (Source: https://www.vidal.ru/drugs/phlebodia_600__4622; accessed: September 4, 2023).

   Diosmin 600 dosing regimen is 600 mg once daily for 2 months.
3. Hesperidin + Diosmin 1000. Manufacturer: ALLIUM (Russia). Active substance: diosmin and hesperidin.

A venotonic agent that also has angioprotective properties. It reduces venous distensibility and blood stasis, reduces capillary permeability and increases their resistance. The results of clinical studies confirm the pharmacological activity of drugs containing this active substance in relation to the parameters of venous hemodynamics. It increases venous tone: a reduction in the time of venous emptying has been demonstrated in studies with venous occlusion plethysmography. In patients with signs of severe microcirculatory disorders the treatment with drugs containing this active substance is associated with a statistically significant (as compared to placebo) improvement in the capillary resistance, which has been proven by angiostereometry. The drug has a proven efficacy in the treatment of CVD of the lower extremities (Source: https://www.vidal.ru/drugs/gesperidin-diosmin; accessed: September 4, 2023).

Hesperidin + Diosmin 1000 dosing regimen is 1000 mg once daily for 2 months. All three of these drugs are venotonic and venoprotective drugs used in the CVD treatment. They are comparable in their pharmacological properties, product labels, profile of side effects and adverse events, and the cost per package of 30 tablets, according to the Moscow chain of pharmacies (Source: https://gorzdrav.org/p/detraleks-tabl-p-o-1000mg-n30-62440/; https://gorzdrav.org/p/flebodia-600-tabl-p-o-600mg-n30-17602/; https://gorzdrav.org/p/venarus-tabl-p-o-900mg-100mg-n30-64844/; accessed: September 4, 2023).

Patients will take these VADs at the same time every morning, during breakfast. Patients will be warned in advance about possible side effects and adverse events. In a case of their occurrence, the patients shall immediately notify the principal investigator or investigators using one or more mobile phone numbers provided to them in advance.

Methodology The study will include 150 consecutive female patients with symptomatic PeVD, according to the inclusion/non-inclusion criteria. All patients will undergo a clinical examination, transabdominal and transvaginal DUS of the pelvic veins to verify the diagnosis and to determine the diameters of the pelvic veins and the duration of reflux in them. The study will include patients with PeVD and isolated dilation and reflux in the parametrial and uterine veins. Previous studies have shown that the use of VADs in patients with a combination of reflux in the ovarian, parametrial and uterine veins is ineffective. The CPP intensity will be assessed using a visual analogue scale (VAS), which is a 10-cm horizontal line ranged from 0 to 10 scores (1 cm equals 1 score). The CPP intensity will be assessed by VAS scores as following: 0, no pain; 1-3, mild pain; 4-6, moderate pain; 7-10, severe pain. After a brief instruction by an investigator, the patients will rate their pain intensity by making a mark on the line.

For randomization procedure, the sealed envelope principle will be used. Three groups of 50 patients each will be formed depending on the recommended VAD usage: group 1 (n=50) with MPFF1000; group 2 (n=50) with Diosmin 600; and group 3 (n=50) with Hesperidin + Diosmin 1000. After the start of VAD intake, the patients will be self-rating the pain intensity on VAS on the weekly basis. After 60 days from the VAD treatment start, the patients will undergo repeated clinical examination and provide an investigator with 8 completed VAS forms. Based on the repeated examination data and the VAS results, a comparative analysis of the clinical efficacy of VADs will be carried out. In a case of side effect or adverse event occurrence during a 2-month treatment course, patients inform the doctor-investigator about it within one day, and the decision is made either to continue, change the regimen of treatment or to discontinue it.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 45 years;
* The presence of PeVD symptoms (CPP, dyspareunia, discomfort in the hypogastrium, dysuria, vulvar varicose veins);
* The presence of pelvic varicose veins with reflux in them, according to DUS;
* Pelvic venous reflux (PVR) lasting for greater than 1 s, according to DUS;
* Isolated dilation and reflux in the parametrial and uterine veins, according to DUS;
* Absence of competing abnormalities, accompanied by CPP.

Exclusion Criteria:

* Asymptomatic form of the disease;
* Menopause;
* Pregnancy;
* Post-thrombotic disease;
* Neoplasms;
* Competing diseases with CPP;
* Known hypersensitivity to any of the components of the used VAD.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Severety of the chronic pelvic pain | Every weekly until 8 weeks
  Evaluation of the efficacy of venoactive drug treatment on chronic pelvic pain by using visual analogue scale

SECONDARY OUTCOMES:
Side and adverse effects | during the treatment until 8 weeks
  Assessment of the frequency and type of of side and adverse effects of venoactive drug therapy

CONTACTS AND LOCATIONS:
Overall Officials: Anatoly V Karalkin, MD, PhD, Study Chair — Pirogov Russian National Research Medical University
Locations (1):
- Pirogov Russian National Research Medical University, Moskva, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Martinez-Zapata MJ, Vernooij RW, Simancas-Racines D, Uriona Tuma SM, Stein AT, Moreno Carriles RMM, Vargas E, Bonfill Cosp X. Phlebotonics for venous insufficiency. Cochrane Database Syst Rev. 2020 Nov 3;11(11):CD003229. doi: 10.1002/14651858.CD003229.pub4. PMID 33141449
- [Background] De Maeseneer MG, Kakkos SK, Aherne T, Baekgaard N, Black S, Blomgren L, Giannoukas A, Gohel M, de Graaf R, Hamel-Desnos C, Jawien A, Jaworucka-Kaczorowska A, Lattimer CR, Mosti G, Noppeney T, van Rijn MJ, Stansby G, Esvs Guidelines Committee, Kolh P, Bastos Goncalves F, Chakfe N, Coscas R, de Borst GJ, Dias NV, Hinchliffe RJ, Koncar IB, Lindholt JS, Trimarchi S, Tulamo R, Twine CP, Vermassen F, Wanhainen A, Document Reviewers, Bjorck M, Labropoulos N, Lurie F, Mansilha A, Nyamekye IK, Ramirez Ortega M, Ulloa JH, Urbanek T, van Rij AM, Vuylsteke ME. Editor's Choice - European Society for Vascular Surgery (ESVS) 2022 Clinical Practice Guidelines on the Management of Chronic Venous Disease of the Lower Limbs. Eur J Vasc Endovasc Surg. 2022 Feb;63(2):184-267. doi: 10.1016/j.ejvs.2021.12.024. Epub 2022 Jan 11. No abstract available. PMID 35027279
- [Background] Nicolaides A, Kakkos S, Baekgaard N, Comerota A, de Maeseneer M, Eklof B, Giannoukas AD, Lugli M, Maleti O, Myers K, Nelzen O, Partsch H, Perrin M. Management of chronic venous disorders of the lower limbs. Guidelines According to Scientific Evidence. Part I. Int Angiol. 2018 Jun;37(3):181-254. doi: 10.23736/S0392-9590.18.03999-8. No abstract available. PMID 29871479
- [Background] Antignani PL, Lazarashvili Z, Monedero JL, Ezpeleta SZ, Whiteley MS, Khilnani NM, Meissner MH, Wittens CH, Kurstjens RL, Belova L, Bokuchava M, Elkashishi WT, Jeanneret-Gris C, Geroulakos G, Gianesini S, de Graaf R, Krzanowski M, Al Tarazi L, Tessari L, Wikkeling M. Diagnosis and treatment of pelvic congestion syndrome: UIP consensus document. Int Angiol. 2019 Aug;38(4):265-283. doi: 10.23736/S0392-9590.19.04237-8. Epub 2019 Jul 24. No abstract available. PMID 31345010
- [Background] Simsek M, Burak F, Taskin O. Effects of micronized purified flavonoid fraction (Daflon) on pelvic pain in women with laparoscopically diagnosed pelvic congestion syndrome: a randomized crossover trial. Clin Exp Obstet Gynecol. 2007;34(2):96-8. PMID 17629162
- [Background] Akhmetzianov RV, Bredikhin RA. Clinical Efficacy of Conservative Treatment with Micronized Purified Flavonoid Fraction in Female Patients with Pelvic Congestion Syndrome. Pain Ther. 2021 Dec;10(2):1567-1578. doi: 10.1007/s40122-021-00312-6. Epub 2021 Sep 19. PMID 34537951
- [Background] Gavrilov SG, Moskalenko YP, Karalkin AV. Effectiveness and safety of micronized purified flavonoid fraction for the treatment of concomitant varicose veins of the pelvis and lower extremities. Curr Med Res Opin. 2019 Jun;35(6):1019-1026. doi: 10.1080/03007995.2018.1552043. Epub 2018 Dec 20. PMID 30468077
- [Derived] Gavrilov SG, Moskalenko YP, Grishenkova AS, Chubchenko SV. Venoactive drug treatment for patients with pelvic varicose veins: Results of the single-center, randomized, open-label study (VENOTREAT). Vasc Med. 2025 Oct;30(5):590-598. doi: 10.1177/1358863X251362200. Epub 2025 Aug 25. PMID 40855727
- See also: General information about micronized purified flavonoid fraction 1000 — https://www.vidal.ru/drugs/detralex__38634
- See also: General information about Diosmin 600 — https://www.vidal.ru/drugs/phlebodia_600__4622

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2024-09-03): https://cdn.clinicaltrials.gov/large-docs/99/NCT06584799/Prot_ICF_001.pdf